CLINICAL TRIAL: NCT00651274
Title: A Multicenter, Randomized, Parallel Groups, Placebo-Controlled Study Comparing The Efficacy, Safety, And Tolerability Of The Daily Co-administration Of Ezetimibe 10 Mg Or Ezetimibe Placebo To Ongoing Treatment With Simvastatin 20 Mg In Subjects With Primary Hypercholesterolemia And Coronary Heart Disease
Brief Title: Comparison of Co-administration of Ezetimibe Plus Simvastatin Versus Simvastatin Alone in Primary Hypercholesterolemia (P03476)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03476
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerosis; Hypercholesterolemia; Coronary Heart Disease
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Experimental)
  Interventions: Drug: Ezetimibe
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe — oral tablets: ezetimibe 10 mg once daily for 6 weeks (plus continued simvastatin)
  Other Names: SCH 58235
  Arms: Ezetimibe
Drug: Placebo — oral tablets: placebo to match ezetimibe 10 mg once daily for 6 weeks (plus continued simvastatin)
  Arms: Placebo

SUMMARY:
This study will assess whether the daily co-administration of ezetimibe 10 mg with ongoing treatment of simvastatin 20 mg will be more effective than treatment with simvastatin 20 mg alone in further reducing LDL-C concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >= 18 years and <= 75 years of age.
* Subjects must have an LDL-C concentration >= 2.6 mmol/L (100 mg/dL) to <= 4.1 mmol/L (160 mg/dL) using the Friedewald calculation available at the time of randomization Visit 3 (Baseline Visit).
* Subjects must have triglyceride concentrations of < 3.99 mmol/L (350 mg/dL) at Visit 3 (Baseline Visit).
* Subjects must have documented coronary heart disease (CHD). For the purposes of this study, CHD will include one or more of the following features: documented stable angina (with evidence of ischemia on exercise testing); history of myocardial infarction; history of percutaneous coronary intervention (primarily PTCA with or without stent placement); symptomatic peripheral vascular disease (claudication); documented history of atherothrombotic cerebrovascular disease; and/or documented history of unstable angina or non-Q wave myocardial infarction.
* Subject must be currently taking simvastatin 20 mg daily and by history has taken 80% of daily evening doses for the preceding 6 weeks prior to Visit 3 (Baseline Visit).
* Subjects must have liver transaminases (ALT, AST) < 50% above the upper limit of normal, with no active liver disease, and CK < 50% above the upper limit of normal at Visit 3 (Baseline Visit).
* Clinical laboratory tests (CBC, blood chemistries, urinalysis) must be within normal limits or clinically acceptable to the investigator at Visit 3 (Baseline Visit).
* Subjects must have maintained a cholesterol lowering diet program for at least 4 weeks prior to the study and be willing to continue the same diet program during the study.
* Subjects must report a stable weight history for at least 4 weeks prior to entry into study at Visit 3 (Baseline Visit).
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant diseases other than hyperlipidemia or coronary heart disease that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and must agree to remain on their cholesterol-lowering diet and their exercise regimen for the duration of the study.

Exclusion Criteria:

* Subjects whose body mass index (BMI) is >= 30 Kg/m^2 at Visit 3 (Baseline Visit).
* Subjects who consume > 14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2004-08-01 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-cholesterol with ezetimibe added to simvastatin versus continued simvastatin alone. | 6 weeks

SECONDARY OUTCOMES:
Percentage of subjects who achieve target LDL-C as defined by the ESC or NCEP guidelines with ezetimibe added to simvastatin versus continued simvastatin alone | 6 weeks
Percent change from baseline in total cholesterol, HDL-C and triglycerides with ezetimibe added to simvastatin versus continued simvastatin alone. | 6 weeks

REFERENCES:
- [Result] Zubaid M, Shakir DK, Bazargani N, Binbrek A, Gopal R, Al-Tamimi O, Bakir S. Effect of ezetimibe coadministration with simvastatin in a Middle Eastern population: a prospective, multicentre, randomized, double-blind, placebo-controlled trial. J Cardiovasc Med (Hagerstown). 2008 Jul;9(7):688-93. doi: 10.2459/JCM.0b013e3282f3a1b1. PMID 18545068